CLINICAL TRIAL: NCT06791018
Title: Cancer Exercise: A Pragmatic Randomized Controlled Trial Evaluating a Mobile Application in Breast Cancer Survivors.
Brief Title: Cancer Exercise: Evaluation of a Mobile App in Breast Cancer Survivors
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alberta (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: HREBA.CC-24-0455
Record Dates: First submitted 2025-01-14; First posted 2025-01-24 (Actual); Last update posted 2026-01-30 (Actual); Status verified 2026-01

CONDITIONS: Breast Cancer; Breast Cancer Early Stage Breast Cancer (Stage 1-3)
Keywords: Breast neoplasm; Digital technology; Mobile app; Exercise; Behavior
MeSH Terms: conditions — Breast Neoplasms; Motor Activity; Behavior | interventions — Exercise

STUDY DESIGN:
Intervention Model Description: The intervention is a cancer-specific mobile application with the aim of increasing exercise levels in cancer survivors.
Masking Description: Participants and investigators will not be blinded to group assignment given the nature of the intervention.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cancer-specific exercise app (Experimental): Participants randomized in this group will be asked to use the app for 12 weeks. Participants will be ask to preferably spread each exercise session over different days of the week. While exercise equipment is not required, the app includes options for using elastic resistance bands or dumbbells. Following baseline assessment and randomization, participants in the intervention group will receive a brief instructional video on how to download and use the app, along with access to a website offering support materials, guidelines, and additional instructional videos. All participants will complete questionnaires at baseline, 12 weeks (post-intervention), and 3 months follow-up.
  Interventions: Other: Exercise
- Usual care (No Intervention): This group will received the ACSM exercise guidelines.

INTERVENTIONS:
Other: Exercise — Participants will be asked to use a cancer-specific exercise mobile app for 12 weeks. The program is designed to achieve the goal of exercising for at least 90 minutes per week, including aerobic exercise three times a week and resistance training twice a week. While exercise equipment is not required, the app supports the optional use of an elastic resistance band or a pair of dumbbells. The app comes with various features to support the exercise journey. Participants will be able to track their progress through periodic testing, access a library of resources that includes information on exercise, and log any additional workouts they perform outside the app. The exercise prescription will be tailored to daily fatigue levels that will be rated before each workout. This ensures that the program is customized to meet individual needs and abilities.
  Other Names: Cancer-specific exercise app
  Arms: Cancer-specific exercise app

SUMMARY:
This study will examine whether a mobile app increases exercise levels in breast cancer survivors after treatments, reduces fatigue, and improves physical functions. This experimental study has 200 participants placed into one of two groups. One group will be asked to use the cancer-specific exercise app over 12 weeks, and the other group will receive the cancer exercise guidelines. Exercise will be measured by self-report questionnaires before and after the intervention and three months later. Self-report questionnaires will measure fatigue and quality of life. This research will determine whether a simple mobile app helps increase exercise in breast cancer survivors. Mobile apps to increase exercise may be provided to all breast cancer survivors after treatments to help them recover and possibly improve survival.

DETAILED DESCRIPTION:
Exercise is beneficial for breast cancer survivors in alleviating treatment side effects, improving quality of life, and possibly survival. Exercise guidelines for cancer survivors recommend 150 minutes of moderate-intensity or 75 minutes of vigorous-intensity aerobic exercise per week and two days of resistance training. However, the number of breast cancer survivors meeting those guidelines declines during treatments because of symptoms such as fatigue, depression, muscle loss, and treatment toxicity. Mobile applications (apps) are promising tools with the potential to overcome barriers to exercise, such as cost, accessibility, time, and travel, which may reduce social health inequalities. Distanced-based interventions, including mobile apps, yield noteworthy results with favorable responses from cancer survivors. However, the literature provides few details regarding the content and features of mobile apps, hindering the understanding of the potential benefits for cancer survivors. The mobile app Cancer Exercise, developed based on Social-Cognitive Theory incorporating several evidence-based behavior change techniques, has been freely available to cancer survivors since 2020. No study to date has examined the efficacy of any existing mobile app for increasing exercise levels and improving outcomes of breast cancer survivors.

The primary aim of this study is to test the efficacy of the mobile app compared to usual care in increasing exercise levels in breast cancer survivors. The secondary aims are to (1) test the efficacy of the app for reducing fatigue and improving quality of life and physical function, (2) examine the effects of the app on motivation, and (3) determine if the app performs differently in diverse subgroups based on demographic (e.g., age, education, ethnicity, and geography) and clinical variables (e.g., disease stage, previous treatments). It was hypothesized that, compared to usual care, the Cancer Exercise app would improve exercise, fatigue, quality of life, physical function, and motivation, similarly across diverse subgroups.

Individuals diagnosed with stage I-III breast cancer (n=200) will be recruited through the Alberta Cancer Registry and randomly assigned to the app intervention (n=100) or usual care (n=100) receiving exercise guidelines. The goal of the intervention group will be to perform at least 90 minutes of aerobic exercise and two days of resistance exercise per week over 12 weeks. Exercise will be measured the Godin Leisure-Time Exercise Questionnaire at baseline, 12 weeks, and 6 months. The European Organization for Research and Treatment of Cancer (EORTC) core 30-item questionnaire (QLQ-C30) will measure quality of life. Analysis of covariance will compare outcomes between groups while adjusting for important demographic and clinical variables. Interactions (subgroup analysis) involving demographic and clinical variables will also be explored.

This research will provide the first evidence of the efficacy of a mobile app for increasing exercise in breast cancer survivors. The results will contribute to regulation in designing app-based exercise interventions to minimize the potential risk of injury and adverse outcomes for breast cancer survivors. With an effective and tested mobile app, healthcare providers may leverage this resource to facilitate safe and easy exercise referrals for patients.

ELIGIBILITY:
Inclusion Criteria:

* ≥ 18 years of age, diagnosed with histologically confirmed stage I, II, or III breast cancer, > 1 to 5 years after diagnosis (2020-2024) and completed all treatments except hormone therapy, own a smartphone (Apple or Android), able to read and understand English, and interested in increasing exercise.

Exclusion Criteria:

* Not being medically cleared to participate in the exercise intervention by a certified exercise physiologist using the Physical Activity Readiness Questionnaire for Everyone (PAR-Q+) (e.g., known cardiac disease or uncontrolled hypertension), evidence of cancer recurrence, stage IV metastatic breast cancer and unable to walk without material or physical support.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2025-05-23 (Actual); Primary Completion 2025-12-20 (Actual); Study Completion 2026-05-20 (Estimated)

PRIMARY OUTCOMES:
Exercise Level | At baseline (enrollment), 12 weeks (post-intervention), and 3-month follow-up.
  An increase in time in moderate to vigorous exercise levels in minutes per week is the primary endpoint of this study. The efficacy of the app intervention will be assessed by the modified Leisure Score Index from the Godin Leisure-Time Exercise Questionnaire. Participants will be asked to recall their average weekly frequency and duration of light, moderate, and vigorous exercise during the past month that lasted at least 10 minutes and was done during free time. Exercise minutes/week will be calculated for moderate and vigorous exercise. Total exercise minutes will be calculated by adding aerobic minutes and strength minutes.

SECONDARY OUTCOMES:
Health-related quality of life (HRQoL) | At baseline (enrollment), 12 weeks (post-intervention), and 3-month follow-up.
  Assessment of health-related quality of life (HRQoL) using the European Organization for Research and Treatment of Cancer (EORTC) core 30-item questionnaire (QLQ-C30) version 3.0.
  The QLQ-C30 is composed of both multi-item scales and single-item measures. These include five functional scales, three symptom scales, a global health status / quality of life scale, and six single items.
  All of the scales and single-item measures range in score from 0 to 100. A high scale score represents a higher response level.
Cancer-Related Fatigue | At baseline (enrollment), 12 weeks (post-intervention), and 3-month follow-up.
  Cancer-related fatigue will be assessed using the validated Functional Assessment of Cancer Therapy-Fatigue (FACT-F) sub-scale, a 13-item self-report instrument designed to measure fatigue and anemia-related concerns in individuals with cancer. Scores on the Fatigue Subscale range from 0 to 52, with higher scores indicating worse fatigue.
  Fatigue will also be collected dynamically through the app as a just-in-time variable. Participants will self-report their fatigue levels using a scale of 0 to 10, where higher scores indicate greater fatigue. These app-reported measures will provide intra-individual data on fatigue fluctuations over time.
Upper Limb Function | At baseline (enrollment), 12 weeks (post-intervention), and 3-month follow-up.
  The self-reported Disabilities of the Arm, Shoulder, and Hand (DASH) questionnaire will measure upper limb function. The DASH is a 30-item questionnaire with a 5-point Likert scale for each item, producing a score that ranges from 0 to 100. Higher scores indicate greater disability or worse upper limb function. The DASH will be assessed at baseline, post-intervention (12 weeks), and 3-month follow-up.
Exercise behavior | At baseline (enrollment), 12 weeks (post-intervention), and 3-month follow-up.
  Exercise behavior will be assessed using the Capability, Opportunity, Motivation (COM) 6-item questionnaire developed by Keyworth et al. (2020), based on the COM-Behavior (COM-B) model framework. Participants will answer questions about factors influencing exercise behavior, such as support, accessibility, and facilities. Each question will be scored on a 5-point Likert scale ranging from 1 (strongly disagree) to 5 (strongly agree), with higher scores indicating better exercise behavior. The total score will reflect the overall exercise behavior of breast cancer survivors.
Capability for Exercise | At baseline (enrollment), 12 weeks (post-intervention), and 3-month follow-up.
  Capability for exercise will be assessed using the physical and psychological capability subdomains of the COM 6-item questionnaire developed by Keyworth et al. (2020).
  Each question will be scored on a 5-point Likert scale ranging from 1 (strongly disagree) to 5 (strongly agree), with higher scores indicating greater capability.
Opportunity for Exercise | At baseline (enrollment), 12 weeks (post-intervention), and 3-month follow-up.
  Opportunity for exercise will be assessed using the physical and social opportunity subdomains of the COM 6-item questionnaire developed by Keyworth et al. (2020).
  Each question will be scored on a 5-point Likert scale ranging from 1 (strongly disagree) to 5 (strongly agree), with higher scores indicating greater opportunity.
Motivation for Exercise | At baseline (enrollment), 12 weeks (post-intervention), and 3-month follow-up.
  Motivation for exercise will be assessed using the reflective and automatic motivation subdomains of the COM 6-item questionnaire developed by Keyworth et al. (2020).
  Each question will be scored on a 5-point Likert scale ranging from 1 (strongly disagree) to 5 (strongly agree), with higher scores indicating greater motivation. Data will be collected at baseline, 12 weeks, and 3 months follow-up.
Demographic characteristics | At enrollment
  Demographic data will be collected by self-report at baseline and will include age, marital status, education, family income, number and age of children at home, employment status, geography, and ethnicity. The baseline questionnaire will also collect self-reported medical data and will include comorbidities, stage of breast cancer, date of diagnosis, treatment protocol, type of surgery (lumpectomy or mastectomy), type of treatment, and weeks since surgery.

OTHER OUTCOMES:
Number of App Logins Per Week | From enrollment to up to 12 weeks.
  Adherence will be assessed by tracking the number of logins to the mobile app. The app's hosting software is programmed to record usage statistics, and the total number of logins will be recorded weekly. Data will be collected over a 12-week intervention period and reported as the average number of logins per week.
Time Spent on the App (Minutes Per Week) | From enrollment to up to 12 weeks.
  Time spent on the mobile app will be measured in minutes per week. The app's hosting software will track the total duration of active app usage each week. Data will be collected weekly over a 12-week intervention period and reported as the average time spent on the app per week.
Session Intervals on the App | From enrollment to up to 12 weeks.
  Session intervals will be measured as the time between consecutive app usage sessions. The app's hosting software will track and calculate these intervals. Data will be collected weekly over a 12-week intervention period and reported as the average session interval in minutes per day.
Number of participants with exercise intervention-related adverse events | From enrollment through the 12 weeks intervention.
  To evaluate the safety of the exercise program provided in the mobile app, any adverse events during the 12-week intervention will be recorded according to the Common Terminology Criteria for Adverse Events (CTCAE) v4.0. Participants will be informed in the consent form to report any adverse events to the study team via email or phone. Adverse events will be categorized by type (criteria) and grade as indicated by the CTCAE guidelines. Data will be summarized as the number and percentage of participants experiencing adverse events.
User experience and satisfaction with mobile app | ntervention group: post-intervention (12 weeks); Usual Care group: 3-month follow-up
  To assess the app's user experience and satisfaction, participants in the intervention group will complete a post-intervention survey at the 12-week time point. This survey will include questions about overall satisfaction with the app and the usability of its various features and functions. Similarly, participants in the Usual Care group will complete the same survey at their 3-month follow-up.
  After the 12-week intervention, participants in the Usual Care group will be granted access to the app. Satisfaction will be measured using a 5-point Likert scale, with scores ranging from 1 (very dissatisfied) to 5 (very satisfied), with higher scores indicating better satisfaction.

CONTACTS AND LOCATIONS:
Locations (1):
- Exercise Oncology Research Laboratory, Faculty of Kinesiology, Sport and Recreation, University of Alberta., Edmonton, Alberta, Canada

IPD SHARING:
Plan to Share IPD: No